CLINICAL TRIAL: NCT06923124
Title: A Retrospective, Non-interventional, Single-center Study to Describe a Spanish Cohort of Patients With FMF and to Identify Suboptimally Treated Patients With Minimal Disease Activity and Its Impact on HRQoL (Health-Related Quality of Life)
Brief Title: A Study to Describe a Group of Spanish Patients With FMF and to Identify Suboptimally Treated Patients With Minimal Disease Activity and Its Impact on Quality of Life
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CACZ885NES01R
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- FMF Cohort: Spanish patients diagnosed with FMF during childhood from January 2005 to December 2021.

SUMMARY:
A retrospective, non-interventional, single-center study conducted in Spain, based on the collection of data from the medical histories of patients with Familial Mediterranean fever (FMF) diagnosed during childhood from January 2005 to December 2021.

Data from the patients' medical records was collected retrospectively, from the time of diagnosis to the current moment of the patient's enrollment in the study. Patients had a minimum follow-up of 3 months after diagnosis.

ELIGIBILITY:
Inclusion criteria:

1. Patients with FMF clinically and/or genetically diagnosed during childhood according to the site's clinical practice.
2. Patients with at least 3 months of follow-up from the date of diagnosis, at the time of their enrollment in the study.

Exclusion criteria:

1. Patients with autoinflammatory disease excluding FMF.
2. Patients with recurrent fever of another etiology (infectious, tumor or other).

Max Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Number of Patients per Clinical Characteristic Category | Baseline
  Clinical characteristic categories included:
  * Diagnostic criteria of FMF (symptom associated with FMF, without a proven infectious cause, with a recurrent pattern and/or accompanied by a genetic test suggestive of Mediterranean FeVer gene [MEFV])
  * Family history of FMF
  * MEFV genotypes
  * Phenotypes of interleukin-1 (IL-1) mediated autoinflammatory disease
  * Diagnosis prior to FMF
Clinical Characteristic: Time From FMF Diagnosis to Study Inclusion | Baseline
Clinical Characteristic: Time From the Start of Symptomatology to Study Inclusion | Baseline
Clinical Characteristic: Time From the Start of Symptomatology to FMF Diagnosis | Baseline
Clinical Characteristic: Age at the Start of Symptomatology | Baseline
Number of Patients by Symptomatology | Baseline, Month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132
  Symptoms included:
  * Abdominal pain
  * Arthralgia
  * Myalgia
  * Articulatory inflammation
  * Chest pain
  * Rash
  * Fatigue
  * Symptoms compatible with Periodic Fever, Aphthous stomatitis, Pharyngitis and Adenitis (PFAPA)
  * Other
Number of Patients by Characteristics of Relapses (Flares) | Baseline, Month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132
  Relapse characteristics included:
  * Fever: high (> 38C), low (≤ 38C), no fever
  * Relapse frequency (<1 or ≥1 relapse per month for 3 months)
  * Presence of triggers
  * Presence of complications
  * Flare and non-flare related inflammatory markers: C-reactive protein (CRP), serum amyloid A protein (SAA), and erythrocyte sedimentation rate (ESR)
  * Disease remission
Flare and Non-flare Related Inflammatory Marker Levels | Baseline, Month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132
  Inflammatory markers included CRP and SAA.
Flare and Non-flare Related Erythrocyte Sedimentation Rate (ESR) | Baseline, Month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132
Number of Flares per Month Since Last Visit | Baseline, Month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132
Flare Duration Since Last Visit | Baseline, Month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132
Number of Patients With Recurrency of Flares at Diagnosis | Baseline
Number of Patients by Comorbidity | Baseline, Month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132
  Comorbidities included vasculitis, panniculitis, inflammatory bowel disease, psoriasis, celiac disease, autoimmune disease, other inflammatory diseases, juvenile idiopathic arthritis, multiple sclerosis, attention deficit hyperactivity disorder (ADHD), and other.
Number of Patients by Treatment Received Before FMF Diagnosis | Baseline
  Treatments included:
  * Non-steroidal anti-inflammatory drugs (NSAIDs)
  * Corticoids
  * Colchicine
  * Anti-IL-1
  * Other
Number of Patients by Treatment Received At Least Once During the Study | Up to 11 years
  Treatments included:
  * Colchicine
  * Canakinumab
  * Anakinra
  * Corticoids
  * Methotrexate (MTX)
  * Anti-IL-6
  * Anti-tumor necrosis factor (TNF)
Number of Patients by Treatment and Treatment Combinations Used at the end of the Study | Up to 11 years
  Treatments and treatment combinations included:
  * Colchicine
  * Canakinumab
  * Anakinra
  * Corticoids
  * MTX
  * Anti-IL-6
  * Anti-TNF
  * Colchicine / Canakinumab
  * Colchicine / Corticoids
  * Anakinra
  * Canakinumab
  * Colchicine / Anti-TNF
  * Colchicine / MTX / Anti-IL- 6
Number of Patients Using Colchicine With Another Treatment at the end of the Study | Up to 11 years
Number of Patients by First Prescribed Colchicine Dose and Age Group | Up to 11 years
Number of Patients by Colchicine Maximum Global Dose and Age Group | Up to 11 years
Number of Patients With a Change in Colchicine Dose | Up to 11 years
Number of Patients by Reason for Stopping Colchicine Treatment and Age Group | Up to 11 years
Number of Patients by Anti-IL-1 Treatment Used at the end of the Study | Up to 11 years
  Anti-IL-1 treatment included canakinumab and anakinra.
Number of Patients by Anti-IL-1 Dose at the end of the Study | Up to 11 years
Number of Patients With a Change in Anti-IL-1 Dose | Up to 11 years
Number of Patients With a Change in Anti-IL-1 Treatment | Up to 11 years
  Changes in treatment included:
  * Change of treatment to a treatment of the same family (anti-IL-1)
  * Change of treatment to a treatment of another family
Number of Patients by Reason for Stopping Anti-IL-1 Treatment | Up to 11 years

SECONDARY OUTCOMES:
Number of Patients by Last Reported Response to Colchicine Treatment | Up to 11 years
  Responses included:
  * Complete response: absence of clinical manifestations and normal CRP/SAA levels.
  * Partial response: <1 flare/month or persistent high CRP/SAA levels with maximum tolerated dose of colchicine or partial response with unknown frequency.
  * Resistant: ≥1 flare/month or persistent high CRP/SAA levels with maximum tolerated dose of colchicine.
  * Intolerant: intolerance to treatment as reason for stopping colchicine treatment or changing to another treatment.
Time to Achieve Response to Colchicine Treatment | Up to 11 years
  Time to achieve first complete response, complete response, and complete response maintenance were measured.
Number of Patients With Intolerance to Colchicine Treatment | Up to 11 years
Autoinflammatory Disease Activity Index (AIDAI) Score | Up to 11 years
  The AIDAI is an assessment tool used to evaluate the level of disease activity. The AIDAI for FMF includes 7 variables: fever, abdominal pain, chest pain, arthralgia or myalgia, swelling of the joints, skin rash, and pain relief taken. Disease activity scores are calculated from the daily scores collected in a patient diary completed during flares. Fever is scored as 0 (absent) or present (1), with all other clinical variables scored from 0 (absent) to 3 (severe). Pain relief taken is not included in the disease activity score calculation. A higher total score indicates a higher level of disease activity.
  AIDAI was used to assess the association between disease activity and colchicine resistance/intolerance, response to canakinumab treatment, pain, fatigue, and quality of life (absenteeism at school during flares, limitation of physical activity, psychological care, and overall health status).
Autoinflammatory Disease Damage Index (ADDI) Score | Up to 11 years
  The ADDI is an assessment tool used to evaluate the level of damage caused by autoinflammatory disease. It consists of 18 damage items grouped by organ system: reproductive, renal/amyloidosis, developmental, serosal, neurological, ears, ocular and musculoskeletal damage. Each damage item is defined and assigned a score of 1, 2, or 3, with each organ system having a maximum allowed score. A higher total score indicates a higher level of damage.
  ADDI was used to assess the association between disease damage and colchicine resistance/intolerance, response to canakinumab treatment, pain, fatigue, and quality of life (absenteeism at school during flares, limitation of physical activity, psychological care, and overall health status).
Familial Mediterranean Fever 50 (FMF50) Score | Up to 11 years
  The FMF50 is an assessment tool used to evaluate response to treatment for FMF. It consists of 6 items:
  1. Percentage change in the frequency of attacks with the treatment.
  2. Percentage change in the duration of attacks with the treatment.
  3. Patients/parents' global assessment of disease severity.
  4. Physicians' global assessment of disease severity.
  5. Percentage change in arthritis attacks with the treatment.
  6. Percentage change in CRP, ESR, or SAA level with the treatment. An improvement of at least 50% in 5 of the 6 items without worsening in any one item indicates that the patient is responding to treatment.
  FMF50 was used to assess response to canakinumab treatment and the association between response to treatment and colchicine resistance/intolerance, pain, fatigue, and quality of life (absenteeism at school during flares, limitation of physical activity, psychological care, and overall health status).
Number of Patients by Last Response Reported to Anti-IL-1 Treatment During the Study | Up to 11 years
  Responses included:
  * Complete response: absence of clinical manifestations and normal CRP/SAA levels.
  * Incomplete response: persistent febrile episodes or high CRP/SAA levels
  * Partial response: <1 flare/month or persistent high CRP/SAA levels with maximum tolerated dose of colchicine or partial response with unknown frequency.
  * Resistant: ≥1 flare/month or persistent high CRP/SAA levels with maximum tolerated dose of colchicine.
  Anti-IL-1 treatments included canakinumab and anakinra.
Time to Achieve Response to Anti-IL-1 Treatment | Up to 11 years
  Time to achieve complete response and complete response maintenance were measured. Anti-IL-1 treatments included canakinumab and anakinra.
Number of Patients With MEFV Mutation by Treatment Response | Up to 11 years
  Response categories included:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Number of Patients Without MEFV Mutation by Treatment Response | Up to 11 years
  Response categories included:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Number of Patients With Mutation in Other Loci by Treatment Response | Up to 11 years
  Response categories included:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Number of Medical Visits of Patients With Scholar Absenteeism During Flares by Response to Anti-IL-1 Treatment | Up to 11 years
  Anti-IL-1 treatments included canakinumab and anakinra. Responses were categorized as follows:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Number of Medical Visits of Patients With Physical Activity Limitations by Response to Anti-IL-1 Treatment | Up to 11 years
  Anti-IL-1 treatments included canakinumab and anakinra. Responses were categorized as follows:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Number of Medical Visits of Patients Requiring Psychological Care by Response to Anti-IL-1 Treatment | Up to 11 years
  Anti-IL-1 treatments included canakinumab and anakinra. Responses were categorized as follows:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Number of Medical Visits of Patients With Presence of Pain by Response to Anti-IL-1 Treatment | Up to 11 years
  Anti-IL-1 treatments included canakinumab and anakinra. Responses were categorized as follows:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Number of Medical Visits of Patients With Presence of Fatigue by Response to Anti-IL-1 Treatment | Up to 11 years
  Anti-IL-1 treatments included canakinumab and anakinra. Responses were categorized as follows:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Visual Analogue Scale (VAS) Score From Clinician Point of View | Up to 11 years
  Patients' overall state of health was assessed using VAS scoring. The VAS is a straight line with a scale ranging from 0 (worst health) to 10 (best health). The clinician marks a point on the line, scoring how they perceive the patient's overall state of health.
  VAS was used to assess the association between anti-IL-1 treatment response and overall state of health. Anti-IL-1 treatments included canakinumab and anakinra. Treatment response was categorized as follows:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.
Visual Analogue Scale (VAS) Score From Patient Point of View | Up to 11 years
  Patients' overall state of health was assessed using VAS scoring. The VAS is a straight line with a scale ranging from 0 (worst health) to 10 (best health). Patients mark a point on the line, scoring how they perceive their overall state of health.
  VAS was used to assess the association between anti-IL-1 treatment response and overall state of health. Anti-IL-1 treatments included canakinumab and anakinra. Treatment response was categorized as follows:
  * Respondent: without flares and with normal inflammatory markers in the last 3 months.
  * Non-respondent: with flare and/or elevated inflammatory markers in the last 3 months.
  * Partial respondent: did not fulfill some of the criteria for complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States